CLINICAL TRIAL: NCT04322656
Title: Stability of Biometry in Patients With Meibomian Gland Dysfunction
Brief Title: Stability of Biometry in Meibomian Gland Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LPF
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Lipiflow; Meibomian gland dysfunction; Biometry
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of Lipiflow treatment on biometrical outcomes (Active Comparator): One eye of each patient will be treated with Lipiflow
  Interventions: Device: Lipiflow treatment
- Control eye (No Intervention): The contralateral eye will serve as control eye

INTERVENTIONS:
Device: Lipiflow treatment — Patients will be treated on one eye with Lipiflow
  Arms: Effect of Lipiflow treatment on biometrical outcomes

SUMMARY:
Accurate biometry is an essential and indispensable tool in preoperative cataract surgery setting to yield optimal postoperative refractive outcome. However, some recent studies indicate that preoperative biometry is influenced by dry eye disease (DED). Hence, the investigator's study aims to investigate the effect of the therapy of MGD using the Lipiflow® device on the stability of biometry and selection of IOL.

DETAILED DESCRIPTION:
Accurate biometry is an essential and indispensable tool in preoperative cataract surgery setting to yield optimal postoperative refractive outcome. 31 Patients suffering from DED caused by MGD will be selected and allocated randomly to therapy. Patients with pre-existing DED therapy other than lubricants will be excluded. After completing prestudy-screening and baseline visit, Lipiflow® therapy is applied to the study eye. Follow-up visits will be scheduled two weeks and three months after baseline visit. Each visit includes dry eye investigations and IOL calculation by IOLmaster 700 and CSO MS-39. After each study visit an IOL will be theoretically selected.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Evidence of meibomian gland dysfunction
* Meibomian gland secretion score equal or less than 15 (for 15 glands of the lower eye lid) using the meibomian gland evaluator (see below)

Exclusion Criteria:

* Usage of eye drops other than lubricants (e.g. antibiotics, steroids, cyclosporin-A)
* Usage of systemic antibiotic therapy
* Any pathology of the ocular surface except dry eye disease (e.g. corneal scarring, cornea ectasia)
* Ocular surgery within prior 3 months
* Ocular injury within prior 3 months
* Ocular herpes of eye or eyelid within prior 3 months
* Active ocular infection
* Active ocular inflammation or history of chronic, recurrent ocular inflammation within prior 3 months
* Eyelid abnormalities that affect lid function
* Ocular surface abnormality that may compromise corneal integrity
* Pregnancy

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Spherical and toric IOL power selected at baseline and at 3 months visit | 12 months
  The difference between pre- and post-treatment biometrical calculated IOL power will be calculated and compared

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria